CLINICAL TRIAL: NCT01034488
Title: Pharmacodynamics Aspects Of Porcine Heparin Sodium, Produced by Eurofarma, Compared Heparin Sodium, Produced by APP Pharmaceuticasls, in Patients With Chronic Renal Failure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: LAL Clínica Pesquisa e Desenvolvimento Ltda, LAL Clínica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HEPEUR1009; Version 01
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heparin sodium - APP (Active Comparator): 5000UI / mL
  Interventions: Biological: Suine
- Heparin - Eurofarma (Experimental): 5000 UI/ mL
  Interventions: Biological: Suine

INTERVENTIONS:
Biological: Suine — 5000UI /mL
  Arms: Heparin sodium - APP
Biological: Suine — 5000UI/mL
  Arms: Heparin - Eurofarma

SUMMARY:
1. Background: Heparin forms a complex with a plasma protein, antithrombin III (ATIII) is an endogenous anticoagulant. This complex inhibits the formation of thrombin and accelerates its destruction. In addition, heparin and ATIII inactivate other proteases of the coagulation cascade, especially the anti-activated factor X. The outcome of these biochemical actions is the inhibition of the formation and synthesis of activators of the clotting factors that exert critical functions in the genesis of the blood clot. Patients with chronic renal failure (CRF) that make use of hemodialysis need a system of anticoagulation with direct inhibitors of thrombin and / or heparinoids to prevent thrombosis.

   Based on clinical studies, the control of plasma heparin level in patients with CRF is essential. Coagulation tests such as APTT, PT, ChT and evidence of activity of anti-Xa factor to be used as a substrate for protection for those patients undergoing hemodialysis.
2. Objective: Check the non-inferiority clinical, the pharmacodynamic effect and safety in use of the drug heparin of porcine origin, produced by the Laboratory Eurofarma, having as the active comparator drug APP ® Heparin Sodium (heparin - APP Pharmaceuticals) in patients with renal failure who do hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of color or social class;
* Age over 18 years, with good clinical doctor's discretion;
* Patients research that agree to participate in the study and sign the informed consent form (attached);
* Chronic renal failure patients in hemodialysis (3 times per week). chronic renal failure patients with indication for anticoagulation during dialysis

Exclusion Criteria:

* Non compliance with the terms described in the informed consent FICT;
* Patients suffering from sensitivity studies heparin sodium;
* Patients with hypersensitivity to search benzyl alcohol;
* Patients with search history of bleeding disorders or disease that a bleeding disorder can worsen or terminate the clinical picture, for example, frames of gastric ulcer;
* Patients with a history of research peptic ulcer;
* Patient with cancer research because of the possibility of impairment of variable coagulation function;
* Patients who are research during pregnancy and postpartum;
* Individuals with a genetic abnormality of the coagulation system;
* Trauma patients;
* Patients on glucocorticoid therapy for at least 1 month;
* Patients using other anticoagulants;
* Patients with a high rate of bleeding;
* Patients undergoing any surgery performed less than 15 days due to the risk of bruising at the site of surgery.
* Patients using drugs that affect hemostasis
* Patients using the following drugs: Salicylates systemic aspirin and other NSAIDs, including ketorolac, Dextran 40, ticlopidine and clopidogrel, systemic glucocorticoids, thrombolytic agents and anticoagulants and other antiplatelet agents, including antagonists of glycoprotein IIb / IIIa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Effect (activity) of heparin observed for markers for aPTT and anti-Xa. | 12 hemodialysis sessions in a row. The sessions take place 3 times a week. So be 4 weeks.

SECONDARY OUTCOMES:
Effectiveness in maintaining the absence clotting during hemodialysis. | 12 consecutive sessions
Safety in use of the drug by monitoring events complicating the use of heparin | 12 consecutive sessions